CLINICAL TRIAL: NCT04435119
Title: COvid-19 et VITamine d en EHPAD
Brief Title: Covid-19 and Vitamin D in Nursing-home
Acronym: COVIT-EHPAD
Status: Completed | Type: Observational
Sponsor: University Hospital, Angers (Other Government)
Responsible Party: Sponsor
Other Study IDs: 2020/67
Record Dates: First submitted 2020-06-12; First posted 2020-06-17 (Actual); Last update posted 2020-06-17 (Actual); Status verified 2020-06

CONDITIONS: Coronavirus
MeSH Terms: conditions — Coronavirus Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
First epidemiological data about COVID-19 pandemic confirm that older adults are likely to experience severe and lethal forms of SARS-CoV-2 infection, in particular frail elderly living in nursing-homes. Vitamin D could be a biological determinant of COVID-19, as indicated by genomic-guided tracing of SARS-CoV-2 targets in human cells. Epidemiological observational data are necessary for better understanding the links between vitamin D supplementation and COVID-19 outcomes, in particular in nursing-homes (in which the risk of hypovitaminosis D is very high).

The investigators had the opportunity to use information collected in a French middle-sized nursing-home affected by COVID-19 in March-April 2020, to determine whether recent vitamin D3 supplementation was associated with the prognosis of COVID-19 in residents infected with SARS-CoV-2. As recommended in French nursing-homes, all residents are systematically and regularly supplemented with bolus vitamin D3 (every single, 2 or 3 months, depending on residents).

The main objective of this study is to determine whether bolus vitamin D3 supplementation taken during or in the month before COVID-19 was effective in improving survival among frail elderly nursing-home residents infected with COVID-19 compared to those having received supplementation longer ago.

The secondary objective is to determine whether bolus vitamin D3 supplementation taken during or in the month before COVID-19 was effective in limiting the clinical severity of the infection according to the World Health Organization's Ordinal Scale for Clinical Improvement (OSCI) for COVID-19 compared to those having received supplementation longer ago.

DETAILED DESCRIPTION:
Retrospective observational unicentric study in nursing-home residents with COVID-19. Health status monitoring data available until May 15, 2020. For all participants, gender, age, disability, history and comorbidities, treatments, date of last vitamin D3 supplementation, results of last blood test, date of suspicion / diagnosis of COVID-19, COVID-19 OSCI score, and eventual hospitalization or death (surveillance data available until May 15, 2020) are collected.

ELIGIBILITY:
Inclusion Criteria:

* Living in the nursing-home of Saint Laurent-de-Chamousset, France, during the COVID-19 epidemic (March-April 2020)
* Being suspected or diagnosed with COVID-19 (RT-PCR, chest CT scan)

Exclusion Criteria:

- Opposition of the resident and/or relatives to the use of anonymized clinical-biological data

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: All residents in the nursing-home of Saint Laurent-de-Chamousset, France, during the COVID-19 epidemic (March-April 2020) This residents are suspected or diagnosed with COVID-19 (RT-PCR, chest CT scan)
Sampling Method: Probability Sample
Enrollment: 96 (Actual)
Dates: Start 2020-03-15 (Actual); Primary Completion 2020-05-15 (Actual); Study Completion 2020-05-15 (Actual)

PRIMARY OUTCOMES:
Number of deaths of any cause in nursing-home residents with SARS-CoV-2 infection, depending on the use of bolus vitamin D3 supplementation during or just before COVID-19 | From March 2020 to 15 May 2020

SECONDARY OUTCOMES:
Clinical severity score of COVID19 in nursing-home residents with SARS-CoV-2 infection, depending on the use of bolus vitamin D3 supplementation during or just before COVID-19 | From March 2020 to 15 May 2020
  Clinical severity score of COVID19 is assessed with Ordinal Scale for Clinical Improvement (OSCI). OSCI ranges from 0 to 8, higher score meaning poorer outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Cédric ANNWEILER, MD, PhD, Principal Investigator — University Hospital, Angers
Locations (1):
- Angers University Hospital, Angers, France